CLINICAL TRIAL: NCT03984097
Title: An Open-Label, Multicenter Phase 1b Study Investigating the Safety of TAK-079 in Combination With Backbone Regimens for the Treatment of Patients With Newly Diagnosed Multiple Myeloma and for Whom Stem Cell Transplantation Is Not Planned as Initial Therapy
Brief Title: A Study to Evaluate Subcutaneous TAK-079 Added to Standard of Care Regimens in Participants With Newly Diagnosed Multiple Myeloma (NDMM)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAK-079-1002; U1111-1230-4820 (Registry Identifier: WHO)
Record Dates: First submitted 2019-06-11; First posted 2019-06-12 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy; TAK-079; CD38; Monoclonal Antibody; Lenalidomide; Bortezomib; Pomalidomide; Velcade; Stem Cell Transplant; Neoplasms, Plasma Cell
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Lenalidomide; Dexamethasone; Bortezomib; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment Phase: TAK-079 and LenDex (Experimental): TAK-079, subcutaneously, once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter, along with lenalidomide, orally, once daily for 21 days and dexamethasone, orally or intravenously, once on Days 1, 8, 15 and 22 in each 28-day treatment until progressive disease (PD) or unacceptable toxicity, withdrawal of consent, death, or termination of the study by sponsor for up to 2 years. The dosage of dexamethasone can be reduced for participants who are greater than (>) 75 years, have poorly controlled diabetes, or had prior intolerance to or AE from corticosteroid therapy.
  Interventions: Drug: TAK-079; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Pomalidomide
- Treatment Phase: TAK-079 and VRd (Experimental): TAK-079 subcutaneously, once weekly for 8 weeks, then once every 2 weeks for 16 weeks, and then once every 4 weeks thereafter, along with bortezomib, subcutaneously, once on Days 1, 8, and 15, for a maximum of 8 cycles, lenalidomide, orally, once daily for 21 days, and dexamethasone, orally or intravenously, once on Days 1, 8, 15 and 22 in each 28-day treatment until PD or unacceptable toxicity, withdrawal of consent, death, or termination of the study by sponsor for up to 2 years. The dosage of dexamethasone can be reduced for participants who are >75 years, have poorly controlled diabetes, or had prior intolerance to or AE from corticosteroid therapy.
  Interventions: Drug: TAK-079; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Bortezomib; Drug: Pomalidomide
- Safety Extension Phase: TAK-079 and, if applicable, backbone therapy (LenDex, VRd, or PomDex) (Experimental): TAK-079 dosing and, if applicable, backbone therapy will be administered as per the schedule outlined in the parent study.
  Interventions: Drug: TAK-079; Drug: Lenalidomide; Drug: Dexamethasone; Drug: Bortezomib; Drug: Pomalidomide

INTERVENTIONS:
Drug: TAK-079 — TAK-079 subcutaneously.
  Other Names: Mezagitamab
Drug: Lenalidomide — Lenalidomide orally.
Drug: Dexamethasone — Dexamethasone orally.
Drug: Bortezomib — Bortezomib subcutaneously.
  Arms: Safety Extension Phase: TAK-079 and, if applicable, backbone therapy (LenDex, VRd, or PomDex); Treatment Phase: TAK-079 and VRd
Drug: Pomalidomide — Pomalidomide orally.

SUMMARY:
The purpose of this original study is to determine the recommended phase 2 dose (RP2D) of TAK-079 when administered to participants with NDMM in combination with the backbone treatment regimen. The purpose of the safety/access cohort is to provide continued access to TAK-079 to participants previously enrolled to a TAK-079 parent study and to evaluate the long-term safety profile of TAK-079.

DETAILED DESCRIPTION:
Treatment phase drug being tested in this study is called TAK-079. TAK-079 is being tested to evaluate the safety, tolerability, efficacy, and pharmacokinetic (PK) when added to 1 of 2 standard backbone regimens (LenDex or VRd) with newly diagnosed NDMM for whom stem cell transplantation (SCT) is not planned as initial therapy.

The study will enroll approximately 36 participants. Participants will be non-randomly assigned to one of the two treatment groups in the original study or Treatment Phase:

* TAK-079 and LenDex
* TAK-079 and VRd

All enrolled participants will have the opportunity to complete the treatment therapy and then enter the Extension study for as long as participants continue to derive benefit. Safety Extension Phase participants who have previously received and tolerated TAK-079-based parent study will continue to the extension study. The study will also evaluate the long-term safety profile of TAK-079. Participants will continue to receive TAK-079 and, if applicable, SOC backbone therapy as per the parent study.

ELIGIBILITY:
Inclusion (Inc) Criteria:

1. Must have previously untreated multiple myeloma (MM) as defined by the IMWG criteria requiring treatment according to the investigator.
2. Are appropriate candidates for either the VRd or Rd backbone antimyeloma therapy according to the investigator.
3. Must have measurable disease defined by at least 1 of the following:

   * Serum M-protein >=1 gram per deciliter (g/dL) (>=10 gram/liter [g/L]).
   * Urine M-protein >=200 mg/24 hours.
   * Serum FLC assay: involved FLC level >=10 mg/dL (>=100 milligram per liter [mg/L]) provided the serum FLC ratio is abnormal.
4. Participants receiving lenalidomide must be able to take concurrent prophylactic anticoagulation per standard clinical practice as directed by the investigator.
5. Life expectancy >3 months.
6. Eastern Cooperative Oncology Group (ECOG) performance status score less than or equal to (<=) 2.

Inc Criteria for Participants in the Safety/Access Cohort (only):

Participants previously treated with TAK-079 therapy in a Takeda-sponsored TAK-079 parent study. Participants will be eligible to enter this cohort when:

1. The parent study is closed, planned to be closed, or has met its primary objectives.

Exclusion (Exc) Criteria:

1. Prior systemic therapy for MM.

   o treatment with bisphosphonates or a single course of glucocorticoids does not disqualify the participant (the maximum dose of corticosteroids should not exceed the equivalent of 160 mg [for example, 40 milligram per day (mg/d) for 4 days] of dexamethasone).
2. Current participation in another interventional study, including other clinical trials with investigational agents (including investigational vaccines or investigational medical device) within 4 weeks of the first dose of TAK-079 or any agent in the backbone regimen and throughout the duration of this trial.
3. Prior radiation therapy within 14 days of the first dose of TAK-079 or any backbone regimen agents.

   NOTE: Prophylactic localized ("spot") radiation for areas of pain is allowed.
4. Major surgery within 4 weeks before Cycle 1 Day 1 (kyphoplasty is not considered major surgery). Participants should be fully recovered from any surgically related complications.
5. Plasmapheresis within 28 days of randomization.
6. If plasmacytoma is the only measurable parameter for assessing disease response, participant is not eligible because of difficult response evaluation.
7. Clinical signs of meningeal involvement of MM exhibited during screening.
8. Serum positive for human immunodeficiency virus (HIV) or active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection.
9. Known severe allergic or anaphylactic reactions to human recombinant proteins or excipients used in the TAK-079 formulation or agents in the backbone regimen (lenalidomide, bortezomib, dexamethasone) as per the respective prescribing information or for TAK-079, as outlined in the current investigator's brochure (IB).
10. Systemic infection requiring systemic antibiotic therapy or other serious infection within 14 days before the first dose of TAK-079 or any agent in the backbone regimen. Urinary tract infection is not considered a systemic infection.
11. A 12-lead electrocardiogram (ECG) showing a QT interval corrected by Frederica's formula (QTcF) >470 milliseconds. If a machine reading is above this value, the ECG should be reviewed by a qualified reader and confirmed on a subsequent ECG.
12. Diagnosis of primary amyloidosis, Waldenstrom's disease, monoclonal gammopathy of undetermined significance (MGUS) or smoldering multiple myeloma (SMM) per IMWG criteria or standard diagnostic criteria, plasma cell leukemia (according to the World Health Organization [WHO] criterion: >=20% of cells in the peripheral blood with an absolute plasma cell count of more than 2 *10^9/L), polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy and skin changes (POEMS syndrome), myelodysplastic syndrome, or myeloproliferative syndrome.
13. History of myelodysplastic syndrome or another malignancy other than MM, except for the following: any malignancy that has been in complete remission for 2 years, adequately treated local basal cell or squamous cell carcinoma of the skin, cervical carcinoma in situ, superficial bladder cancer, asymptomatic prostate cancer (Gleason score <=6 without known metastatic disease and with no requirement for therapy, or requiring only hormonal therapy and stable prostate-specific antigen for >=1 year before initiation of study therapy), breast carcinoma in situ with full surgical resection, and treated medullary or papillary thyroid cancer.

Exc Criteria for Participants in the Safety/Access Cohort

1. Participants meeting any of the criteria for treatment discontinuation in the parent study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-07-29 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Treatment Phase: RP2D of TAK-079 | Up to Cycle 1 (Cycle length is equal to [=] 28 days)
  RP2D of TAK-079 along with lenalidomide-dexamethasone (LenDex) or TAK-079 along with bortezomib, lenalidomide, and dexamethasone (VRd) will be based on number of participants with dose limiting toxicity (DLT). DLTs will be evaluated according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03.
Safety Extension Phase: Number of Participants Reporting one or More Serious Adverse Events (SAEs) | From first dose up to 30 days after the last dose of study drug (up to 4 years)
Safety Extension Phase: Number of Participants With Grade 3 or Higher Treatment-emergent Adverse Events (TEAEs) | From first dose up to 30 days after the last dose of study drug (up to 4 years)
  Adverse event (AE) Grades will be evaluated as per NCI CTCAE, version 4.03.
Safety Extension Phase: Number of Participants Who Require Dose Modification | From first dose up to 30 days after the last dose of study drug (up to 4 years)
Safety Extension Phase: Number of Participants With TEAEs Leading to Treatment Discontinuation | From first dose up to 30 days after the last dose of study drug (up to 4 years)

SECONDARY OUTCOMES:
Treatment Phase: Overall Response Rate (ORR) | Up to 2 years
  ORR based on International Myeloma Working Group (IMWG) Uniform Response Criteria, is defined as the percentage of participants who achieved a PR or better during the study. PR is defined as greater than or equal to (>=) 50 percent (%) reduction of serum M-protein, and reduction in 24-hour urinary M-protein by >=90% or to less than (<) 200 milligram per 24 hours (mg/24 h). If serum and urine M protein are not measurable, >=50% decrease in difference between involved and uninvolved free light chain (FLC) levels is required in place of M protein criteria.
Treatment Phase: Number of Participants Reporting one or More TEAEs and SAEs | From first dose up to 30 days after the last dose of study drug (up to 2 years)
Treatment Phase: Number of Participants With Grade 3 or Higher TEAEs | From first dose up to 30 days after the last dose of study drug (up to 2 years)
  AE Grades will be evaluated as per NCI CTCAE, version 4.03.
Treatment Phase: Number of Participants with TEAEs Leading to Treatment Discontinuation | From first dose up to 30 days after the last dose of study drug (up to 2 years)
Treatment Phase: Number of Participants With AEs Leading to On-study Deaths | From screening up to 30 days after the last dose of study drug (up to 2 years)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (9):
- United States (9):
  - Alabama Oncology, Birmingham, Alabama
  - Pacific Cancer Care, Monterey, California
  - American Oncology Partners of Maryland, PA, Bethesda, Maryland
  - Columbia University Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Good Samaritan Hospital, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f6b603c4db2bf003ab4a340